CLINICAL TRIAL: NCT00296530
Title: A Multicenter, Randomized, Double-Blind, Triple-Dummy, Placebo-Controlled, Parallel Group, Four-Week Study Assessing the Efficacy of Fluticasone Propionate Aqueous Nasal Spray 200mcg QD Versus Montelukast 10mg QD in Adolescent and Adult Subjects With Asthma and Seasonal Allergic Rhinitis Who Are Receiving ADVAIR DISKUS® 100/50mcg BID or Placebo BID
Brief Title: Study Of Patients With Allergic Rhinitis And Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ADA103578
Record Dates: First submitted 2006-02-23; First posted 2006-02-27 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Asthma
Keywords: Asthma; Allergic Rhinitis
MeSH Terms: conditions — Asthma; Rhinitis, Allergic | interventions — Fluticasone-Salmeterol Drug Combination; Fluticasone; montelukast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: fluticasone propionate/salmeterol
Drug: fluticasone propionate
Drug: montelukast
  Other Names: fluticasone propionate/salmeterol; fluticasone propionate

SUMMARY:
This study will last up to 6 weeks. Subjects will visit the clinic up to 5 times. Certain clinic visits will include a physical examination, medical history review, and lung function tests. All study related medications and medical examinations will be provided at no cost to the subject. The drugs used in this study are approved for the age group under study.

DETAILED DESCRIPTION:
A Multicenter, Randomized, Double-Blind, Triple-Dummy, Placebo-Controlled, Parallel Group, Four-Week Study Assessing the Efficacy of Fluticasone Propionate Aqueous Nasal Spray 200mcg QD versus Montelukast 10mg QD in Adolescent and Adult Subjects with Asthma and Seasonal Allergic Rhinitis Who are Receiving ADVAIR DISKUS® 100/50mcg BID or Placebo BID

ELIGIBILITY:
Inclusion Criteria:

* Have asthma for at least 3 months prior to the study.
* Have been using an allowed pre-study asthma therapy for at least 3 months prior to study.
* Currently have seasonal allergic rhinitis and have had seasonal onset of allergic rhinitis for at least the two previous allergy seasons.
* Have a positive allergy skin test.

Exclusion Criteria:

* Have a history of life-threatening asthma.
* Been hospitalized for asthma within the 6 months prior to the study.
* Have certain conditions that would make study participation unsafe.

The study doctor will evaluate other inclusion and exclusion criteria.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2005-09; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Morning Peak Expiratory Flow

SECONDARY OUTCOMES:
Total Nasal Symptom Scores Morning Forced Expiratory Volume in 1 Second Asthma Symptom-Free Days Asthma Rescue-Free Days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (70):
- United States (70):
  - GSK Investigational Site, Ozark, Alabama
  - GSK Investigational Site, Tempe, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, Palmdale, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Jose, California
  - GSK Investigational Site, Stockton, California
  - GSK Investigational Site, Vista, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Wheat Ridge, Colorado
  - GSK Investigational Site, Coral Gables, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Lawrenceville, Georgia
  - GSK Investigational Site, Lilburn, Georgia
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Kenilworth, Illinois
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Covington, Louisiana
  - GSK Investigational Site, Lafayette, Louisiana
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Bethesda, Maryland
  - GSK Investigational Site, Chevy Chase, Maryland
  - GSK Investigational Site, North Andover, Massachusetts
  - GSK Investigational Site, Ypsilanti, Michigan
  - GSK Investigational Site, Rolla, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Ocean City, New Jersey
  - GSK Investigational Site, Skillman, New Jersey
  - GSK Investigational Site, Ithaca, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, North Olmsted, Ohio
  - GSK Investigational Site, Sylvania, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Eugene, Oregon
  - GSK Investigational Site, Lake Oswego, Oregon
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Collegeville, Pennsylvania
  - GSK Investigational Site, Gibsonia, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, East Providence, Rhode Island
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, Germantown, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Corsicana, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, El Paso, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Killeen, Texas
  - GSK Investigational Site, Plano, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Waco, Texas
  - GSK Investigational Site, Murray, Utah
  - GSK Investigational Site, West Jordan, Utah
  - GSK Investigational Site, South Burlington, Vermont
  - GSK Investigational Site, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] This study has not been published in the scientific literature.
- [Derived] Katial RK, Oppenheimer JJ, Ostrom NK, Mosnaim GS, Yancey SW, Waitkus-Edwards KR, Prillaman BA, Ortega HG. Adding montelukast to fluticasone propionate/salmeterol for control of asthma and seasonal allergic rhinitis. Allergy Asthma Proc. 2010 Jan-Feb;31(1):68-75. doi: 10.2500/aap.2010.31.3306. PMID 20167147
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: ADA103578 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: ADA103578 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: ADA103578 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: ADA103578 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: ADA103578 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: ADA103578 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: ADA103578 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register